CLINICAL TRIAL: NCT05522738
Title: Prospective, Single-arm, Single-center Phase Ib/II Trial on the Safety and Efficacy of Fruquintinib in Combination With FOLFIRI in RAS-mutated Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy of Fruquintinib+FOLFIRI in RAS-mutated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Principal Investigator, Dai, Guanghai, Director, Medical Oncology Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-N1-CRC104
Record Dates: First submitted 2022-08-23; First posted 2022-08-31 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: RAS-mutant; second-line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Fruquintinib combined with FOLFIRI
  Interventions: Drug: Combination: Fruquintinib + FOLFIRI

INTERVENTIONS:
Drug: Combination: Fruquintinib + FOLFIRI — Phase 1b Fruquintinib was administered in a 3 + 3 dose escalation regimen at the following doses: L1:3 mg/d, L2:4 mg/d, L3:5 mg/d.
  Fruquintinib: QD po q2w
  FOLFIRI regimen:
  Irinotecan：180 mg/m2, i.v. , d1, q2w LV：200 mg/m2, i.v., d1, q2w 5-FU：2400 mg/m2, i.v.for over 46 hours, q2w
  Phase II Fruquintinib: RP2D, QD po q2w
  FOLFIRI regimen:
  Irinotecan： 180 mg/m2, i.v. , d1, q2w LV： 200 mg/m2, i.v., d1, q2w 5-FU：2400 mg/m2, i.v.for over 46 hours, q2w
  Other Names: Elunate; HMPL-013

SUMMARY:
Molecular subtypes make difference on clinicopathologic features and response to chemotherapy and targeted agents as well as prognosis. RAS mutation status, which accounting for approximately 35% to 40% of colorectal cancer patients, is an important factor considered in the standard of care for colorectal cancer. For RAS-mutated patients, no targeted driver gene drugs have been approved, and their treatment is based on the anti-VEGF/VEGFR pathway, and corresponding targeted drugs such as bevacizumab, aflibercept, and ramucirumab have also been successfully marketed for the treatment of CRC.

For RAS mutant metastatic colorectal cancer, the commonly used first-line treatment regimen is bevacizumab combined with chemotherapy, which is shown in previous studiesthat the PFS of 1st-line is about 10 months; the standard regimen of second-line treatment is FOLFIRI ± bevacizumab, which is shown in previous study that the 2nd-line PFS is about 5 months with ORR 4%. There are a lot of unmet medical needs to improve the clinical efficacy in secondline-treatment of RAS-mutant patients.

DETAILED DESCRIPTION:
This is a prospective, single-armed, single-center phase Ib/II study to investigate the safety and efficacy of Fruquintinib combined with FOLFIRI in RAS-mutant patients who failed first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the study and voluntarily sign the informed consent form;
2. Age ≥ 18 years;
3. Pathologically confirmed unresectable metastatic colorectal cancer;
4. Known RAS gene mutations;
5. failed standard first-line FOLFOX/XELOX combined with bevacizumab;
6. ECOG performance status 0-1;
7. BMI ≥ 18;
8. Expected survival ≥ 3 months;
9. Vital organ function meets the following requirements (any blood components and cell growth factors are not allowed within 14 days before enrollment):

   * Absolute neutrophil count ≥ 1.5 × 109/L and white blood cells ≥ 4.0 × 109/L;
   * Platelets ≥ 100 x 109/L;
   * Hemoglobin ≥ 90 g/L;
   * Total bilirubin TBIL ≤ 1.5 × ULN;
   * ALT and AST ≤ 5 x ULN;
   * Urea nitrogen/urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 x ULN (and creatinine clearance (CCr) ≥ 50 mL/min);
   * Left ventricular ejection fraction (LVEF) > = 50%;
   * Fridericia corrected QT interval (QTcF) < 470 milliseconds.
   * INR ≤ 1.5 x ULN, APTT ≤ 1.5 x ULN.
10. Women of childbearing age should take effective contraceptive measures;
11. Good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Unable to comply with the study protocol or study procedures;
2. Known BRAF gene mutations;
3. evidence of central nervous system metastasis, or associated with severe malignant pleural effusion and ascites;
4. Previous treatment with irinotecan;
5. previous treatment with VEGFR inhibitor
6. Concurrent use of any other investigational drug, or enrollment in a clinical trial of other investigational drug therapy within 4 weeks before enrollment;
7. Inactivated vaccines within 4 weeks before enrollment or possibly during the study;
8. patients in the study group underwent major surgery or severe traumatic injury, fracture or ulcer within 4 weeks;
9. Receiving blood transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony-stimulating factor (G-CSF), within 28 days before enrollment;
10. Alcohol or drug abuse within 4 weeks prior to enrollment;
11. Any factor affecting oral administration;
12. Concurrent any of the following: uncontrolled hypertension, coronary artery disease, arrhythmia, and heart failure;
13. Uncontrollable serious concurrent infections resulting in disability;
14. Proteinuria ≥ 2 + (1.0 g/24 h)
15. Evidence or history of bleeding tendency within 2 months before enrollment, regardless of seriousness;
16. Arterial/venous thromboembolic events, such as cerebrovascular accidents (including transient ischemic attack), within 12 months before the first treatment;
17. Acute myocardial infarction, acute coronary syndrome or CABG within 6 months prior to the first treatment;
18. Fractures or wounds that have not been healed for a long time;
19. Coagulopathy, bleeding tendency, or ongoing anticoagulant therapy;
20. Patients with other malignant tumors within 5 years before enrollment, except for skin basal cell carcinoma or squamous cell carcinoma after radical resection, or cervical carcinoma in situ;
21. Active autoimmune disease or history of autoimmune disease within 4 weeks before enrollment;
22. Previous allogeneic bone marrow transplantation or organ transplantation;
23. Subjects who are allergic to the study drug or any of its excipients;
24. clinically significant electrolyte abnormalities judged by the investigator;
25. Known human immunodeficiency virus (HIV) infection. Known history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must have excluded active HBV infection, ie, positive HBV DNA (> 1 × 104 copies/mL or > 2000 IU/mL); known hepatitis C virus (HCV) infection and positive HCV RNA (> 1 × 103 copies/mL);
26. Unresolved toxicities above CTCAE v5.0 grade 1 due to any prior anticancer therapy, excluding alopecia, lymphopenia, and oxaliplatin-induced neurotoxicity ≤ grade 2;
27. Any other diseases, clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the investigator 's judgment, there is reason to suspect that the patient has a disease or condition that is not suitable for the use of the study drug (such as having seizures and requiring treatment), or will affect the interpretation of the study results, or put the patient at high risk;
28. Pregnant or lactating females;
29. Patients who the investigator considers inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From treatment initiation to progressive disease or EOT due to any cause, assessed up to 1 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
RP2D | from first dose up to progressive disease or EOT due to any cause, assessed up to 1 year
  RECIST v1.1

SECONDARY OUTCOMES:
Overall Survival | from treatment initiation until death due to any cause, assessed up to 3 year
  every two months follow up after EOT observation period at 30 days after the last medication
Progress-Free Survival | from treatment initiation until death due to any cause, assessed up to 2 year
  every two months follow up after EOT observation period at 30 days after the last medication
Duration of Response | from treatment initiation until death due to any cause, assessed up to 2 year
  every two months follow up after EOT observation period at 30 days after the last medication
Safety and tolerance evaluated by incidence of AE | from first dose to 30 days post the last dose
  Incidence and severity of AE
Safety and tolerance evaluated by incidence of SAE | from first dose to 30 days post the last dose
  Incidence and severity of SAE

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Doctor, Principal Investigator — Chinese PLA General Hospital; Quanli Han, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No